CLINICAL TRIAL: NCT03785509
Title: The Effect of Persistence and Compliance of Antiplatelet and Dyslipidemia Agents on Cardiovascular Outcomes in Real World Patients Undergoing Percutaneous Coronary Intervention
Brief Title: The Compliance of DAPT and Statins on Clinical Outcomes in Percutaneous Coronary Intervention Patients
Acronym: CPPCI
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Ho Choi, MD, PhD, Professor, Samsung Medical Center
Other Study IDs: SMC 2017-04-014-001
Record Dates: First submitted 2018-12-16; First posted 2018-12-24 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Platelet Aggregation Inhibitors; Hydroxymethylglutaryl-coa Reductase Inhibitors; Compliance, Medication; Adherence, Medication; Persistence, Medication; Percutaneous Coronary Intervention
Keywords: DAPT, Statin, Compliance, Persistence, Adherence, PCI
MeSH Terms: conditions — Medication Adherence; Patient Compliance | interventions — 2'-deoxythymidylyl-(3'-5')-2'-deoxyadenosine; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: DAPT, Statin — Compliance of DATP, Compliance of Statin, Drug Eluting Stent, Bare Metal Stent
  Other Names: DES, BMS

SUMMARY:
A nationwide retrospective cohort study. To investigate the real world medication compliance and the relation with clinical outcomes.

The persistence and compliance to dual anti-platelet therapy(DAPT) and dyslipidemia agents are important for the patients undergoing percutaneous coronary intervention. But, the discontinuation and compliance rate are unknown in the real world setting.

DETAILED DESCRIPTION:
A nationwide retrospective cohort study. The persistence and compliance to dual anti-platelet therapy(DAPT) and dyslipidemia agents are important for the patients undergoing percutaneous coronary intervention. The discontinuation and uncompliance may increase a risk. But, the discontinuation and compliance rate are not well known in the real world patients undergoing bare metal stents(BMS) and drug eluting stents(DES) insertion.

To investigate the real world medication compliance and the relation with clinical outcomes, administrative claim data was extracted from the Korean National Healthcare Insurance(KNHI) database.

All Korean patient date undergoing PCI from January 1, 2011 to December 2011 is extracted. 5 year clinical outcomes are investigated.

Primary outcomes are the MACE including all-cause death, revascularization, critically ill status, and stroke) classified by the medication compliance. Medication complinace is measured by proportion of days covered(PDC)

Secondary outcomes are the patterns of medication persistence and its outcomes to understand critical points.

ELIGIBILITY:
Inclusion Criteria:

1. All claim of percutaneous coronary intervention using stent in the National Healthcare Insurance Service of Korea between January 1st 2011 and December 31st, 2011

Exclusion Criteria:

1. No use of stents
2. Stent not classified into DES or BMS
3. Use of DES and BMS together at the same initial day

Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing PCI using stents in 2011 from all medical providers in Korea is selected using National Health Insurance Services.
Sampling Method: Non-Probability Sample
Enrollment: 47291 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2018-02-06 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence density of MACE | 5 years
  5 year incidence densities of a major adverse clinical events(MACEs) consisting of all-cause death, revascularization, critically ill status and stroke.

SECONDARY OUTCOMES:
Compliance defined as a proportion of days covered (%) | 6 month
  PDC (Proportion of days covered)

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Ho Choi, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Gang nam-Gu, Ilwon-Dong, South Korea